CLINICAL TRIAL: NCT02876692
Title: Prediction and Management of Delayed Graft Function Based on Donor Criteria and LifePort Platform
Acronym: Xi'anCri
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Principal Investigator, Ding Xiaoming, Director of renal transplant department, First Affiliated Hospital Xi'an Jiaotong University
Other Study IDs: XAC-01
Record Dates: First submitted 2016-08-19; First posted 2016-08-24 (Estimated); Last update posted 2016-09-01 (Estimated); Status verified 2016-08

CONDITIONS: Delayed Graft Function
MeSH Terms: conditions — Delayed Graft Function

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Machine perfusion — Deceased donor kidneys were preserved by hypothermic machine perfusion

SUMMARY:
This is a prospective cohort study:

1. First step: to establish a new scoring system for predication of delayed graft function(DGF) following kidney transplantation based on previous and new study data. The new scoring system is comprised of two parts: Xi'an Criteria of donor scoring system and kidney evaluation System based on Lifeport platform ).
2. Second step: validate the new scoring system through prospective cohort study in our transplantation center and modify the scoring system if needed. Recruiting 300 patients, follow up at day 3, week 1, month 1, month 3, month 6 and month 12. Patients will be followed for Cr30cl, DGF,primary non-function (PNF), acute rejection (AR), graft survival and patient survival
3. Step 3: Further validate the new scoring system in six other transplantation centers and developing a software in the end. Recruiting 300 patients, follow up at day 3, week 1, month 1, month 3, month 6 and month 12. Patients will be followed for Cr30cl, DGF, PGF, AR, graft survival and patient survival

DETAILED DESCRIPTION:
Subjects are enrolled to collect the data of donors and recipients. Investigators also collect the data of recipients or donated organs as following: physiological and biochemical indexes, machine perfusion parameters, and the other factors effected on renal transplant outcomes. A Cox proportional hazards model and multiple linear regression analysis will be applied to examine the correlation among the univariate and multivariate. Based on the above analysis to improve the new scoring system, Lifeport work platform evaluation system and donor kidney quality evaluation system. Then, a multi-center clinical trial will be started to improve and verify the new scoring system. Finally, a donor kidney evaluation APP will be developed based on the scoring system and the database of clinical trials. An applicaiotion (APP) will be popularized the national transplant surgeons.

ELIGIBILITY:
Inclusion Criteria:

Donor

* 1. Comply with the national donation after citizen death guideline
* 2. No high risk activities: such as history of drug abuse, history of intravenous drug use and risky sexual behavior
* 3. No malignant melanoma, metastatic cancer, or incurable cancer; some of the early stages of cancer after a successful treatment can also be considered
* 4. No activity of untreated systemic bacterial, viral or fungal infection;
* 5. Patients definitely identified

Recipient:

* 1. 65 y old ≥Age> = 18 years old, male or female
* 2. BMI<26
* 3. Renal transplantation first time
* 4. Not in pregnancy or lactation, pregnancy test was negative, and promise not to be pregnant during treatment.
* 5. Before the clinical trial, Patient sign informed consent voluntarily

Exclusion Criteria:

Donor

* 1. Older than 65 years old
* 2.Serum hepatitis B virus (HBV), hepatitis C virus (HCV), HIV positive
* 3.Donor kidney cold storage time over 30 hours
* 4.Warm ischemia time over 20 minutes
* 5.Other reagents are added perfusion for regulation of donor renal function

Recipient:

* 1.Involved in other study.
* 2.Double organ or multi-organ transplant
* 3.A,B,O blood type-incompatible

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients assigned the deceased donor kidney to transplant in the waiting list.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2016-01; Primary Completion 2018-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
delayed graft function | 7 days after renal transplant
Transplant nephrectomy | 1 year after reanl transplant

SECONDARY OUTCOMES:
Abnormal serum creatinine | Serum creatinine did not return to the normal range within the first 30 days
Renal dysfunction caused by the acute rejection | within the first 3 months
lung infection lead to death | within the first 1 year
Renal dysfunction caused by Surgical complications | within the first 3 months

CONTACTS AND LOCATIONS:
Overall Officials: xiaoming D Ding, PhD, Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- First Affiliated Hospital Xi'an Jiaotong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Allen AM, Kim WR, Xiong H, Liu J, Stock PG, Lake JR, Chinnakotla S, Snyder JJ, Israni AK, Kasiske BL. Survival of recipients of livers from donation after circulatory death who are relisted and undergo retransplant for graft failure. Am J Transplant. 2014 May;14(5):1120-8. doi: 10.1111/ajt.12700. Epub 2014 Apr 14. PMID 24731165
- [Background] Huang J, Millis JM, Mao Y, Millis MA, Sang X, Zhong S. A pilot programme of organ donation after cardiac death in China. Lancet. 2012 Mar 3;379(9818):862-5. doi: 10.1016/S0140-6736(11)61086-6. Epub 2011 Nov 10. PMID 22078722
- [Background] Huang J, Wang H, Fan ST, Zhao B, Zhang Z, Hao L, Huo F, Liu Y. The national program for deceased organ donation in China. Transplantation. 2013 Jul 15;96(1):5-9. doi: 10.1097/TP.0b013e3182985491. PMID 23743728
- [Background] World Health Organization. WHO guiding principles on human cell, tissue and organ transplantation. Transplantation. 2010 Aug 15;90(3):229-33. doi: 10.1097/TP.0b013e3181ec29f0. No abstract available. PMID 20664493
- [Background] Moers C, Leuvenink HG, Ploeg RJ. Non-heart beating organ donation: overview and future perspectives. Transpl Int. 2007 Jul;20(7):567-75. doi: 10.1111/j.1432-2277.2007.00455.x. Epub 2007 Jan 30. PMID 17263786
- [Background] Kokkinos C, Antcliffe D, Nanidis T, Darzi AW, Tekkis P, Papalois V. Outcome of kidney transplantation from nonheart-beating versus heart-beating cadaveric donors. Transplantation. 2007 May 15;83(9):1193-9. doi: 10.1097/01.tp.0000261710.53848.51. PMID 17496535
- [Background] Jochmans I, Darius T, Kuypers D, Monbaliu D, Goffin E, Mourad M, Ledinh H, Weekers L, Peeters P, Randon C, Bosmans JL, Roeyen G, Abramowicz D, Hoang AD, De Pauw L, Rahmel A, Squifflet JP, Pirenne J. Kidney donation after circulatory death in a country with a high number of brain dead donors: 10-year experience in Belgium. Transpl Int. 2012 Aug;25(8):857-66. doi: 10.1111/j.1432-2277.2012.01510.x. Epub 2012 Jun 13. PMID 22694305
- [Background] Chamorro C, Falcon JA, Michelena JC. Controversial points in organ donor management. Transplant Proc. 2009 Oct;41(8):3473-5. doi: 10.1016/j.transproceed.2009.09.004. PMID 19857774
- [Background] Gelb AW, Robertson KM. Anaesthetic management of the brain dead for organ donation. Can J Anaesth. 1990 Oct;37(7):806-12. doi: 10.1007/BF03006543. PMID 2225301
- [Result] Xue W, Tian P, Ding X, Pan X, Yan H, Hou J, Feng X, Xiang H, Tian X, Ren L, Zheng J, Li S. Clinical research and social status investigation for donor and recipient of living-related kidney transplant. Int Urol Nephrol. 2013 Feb;45(1):239-49. doi: 10.1007/s11255-012-0259-0. Epub 2012 Aug 15. PMID 22893495
- [Result] Wadei HM, Heckman MG, Rawal B, Taner CB, Farahat W, Nur L, Mai ML, Prendergast M, Gonwa TA. Comparison of kidney function between donation after cardiac death and donation after brain death kidney transplantation. Transplantation. 2013 Aug 15;96(3):274-81. doi: 10.1097/TP.0b013e31829807d1. PMID 23778649
- [Result] Singh RP, Farney AC, Rogers J, Zuckerman J, Reeves-Daniel A, Hartmann E, Iskandar S, Adams P, Stratta RJ. Kidney transplantation from donation after cardiac death donors: lack of impact of delayed graft function on post-transplant outcomes. Clin Transplant. 2011 Mar-Apr;25(2):255-64. doi: 10.1111/j.1399-0012.2010.01241.x. PMID 20331689
- [Result] Mallon DH, Summers DM, Bradley JA, Pettigrew GJ. Defining delayed graft function after renal transplantation: simplest is best. Transplantation. 2013 Nov 27;96(10):885-9. doi: 10.1097/TP.0b013e3182a19348. PMID 24056620
- [Result] Nagaraja P, Roberts GW, Stephens M, Horvath S, Fialova J, Chavez R, Asderakis A, Kaposztas Z. Influence of delayed graft function and acute rejection on outcomes after kidney transplantation from donors after cardiac death. Transplantation. 2012 Dec 27;94(12):1218-23. doi: 10.1097/TP.0b013e3182708e30. PMID 23154212
- [Result] Lodhi SA, Lamb KE, Uddin I, Meier-Kriesche HU. Pulsatile pump decreases risk of delayed graft function in kidneys donated after cardiac death. Am J Transplant. 2012 Oct;12(10):2774-80. doi: 10.1111/j.1600-6143.2012.04179.x. Epub 2012 Jul 23. PMID 22823748